CLINICAL TRIAL: NCT02678975
Title: DIRECT (DIsulfiram REsponse as add-on to ChemoTherapy in Recurrent) Glioblastoma: A Randomized Controlled Trial
Brief Title: Disulfiram in Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); Lund University Hospital (Other); Karolinska University Hospital (Other); University Hospital, Linkoeping (Other); Region Örebro County (Other); Ryhov County Hospital (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Asgeir S. Jakola, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: no ID yet
Record Dates: First submitted 2016-01-31; First posted 2016-02-10 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Disulfiram; Copper; Alkylating Agents; Lomustine; Temozolomide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Alkylating chemotherapy
  Interventions: Drug: Alkylating Agents
- Experimental (Experimental): Alkylating chemotherapy + disulfiram + copper
  Interventions: Drug: Disulfiram; Dietary Supplement: Copper; Drug: Alkylating Agents

INTERVENTIONS:
Drug: Disulfiram — Disulfiram 400 mg daily
  Arms: Experimental
Dietary Supplement: Copper — nutritional supplement with copper, 2 mg daily
  Arms: Experimental
Drug: Alkylating Agents — Alkylating antineoplastic agent
  Other Names: lomustine (CCNU), PCV or temozolomide

SUMMARY:
Disulfiram (Antabuse®) is a well-tolerated, cheap, generic drug that has been in use since the 1950s to treat alcoholism. There is now an increasing amount of independent preclinical data to support disulfiram as an anticancer agent. The potency of disulfiram as an anticancer agent seems strengthened by copper.

The investigators aim is to investigate disulfiram and copper-supplement as add-on treatment in glioblastoma patients with recurrence receiving alkylating chemotherapy.

DETAILED DESCRIPTION:
Disulfiram (Antabuse®) is a well-tolerated, cheap, generic drug that has been in use since the 1950s to treat alcoholism. There is now an increasing amount of independent preclinical data to support disulfiram as an anticancer agent. The potency of disulfiram as an anticancer agent seems strengthened by copper. There is now anecdotal clinical evidence of disulfiram as an anticancer agent. So far no clinical studies have been published in glioma patients, but two small, uncontrolled studies are planned according to clinicaltrials.gov. with search 1st November 2015.

The investigators aim to investigate disulfiram and copper-supplement as add-on treatment in glioblastoma patients with recurrence receiving alkylating chemotherapy. The study will be performed as a multicenter RCT including patients in Norway and Sweden. This will serve as a proof-of concept study.

The primary end-point is survival at 6 months

ELIGIBILITY:
Inclusion Criteria:

1. A previous diagnosis of glioblastoma (histologically verified) and presenting with a first progression/recurrence documented by MRI.
2. Indication for treatment with chemotherapeutic alkylating agents (i.e. temozolomide OR lomustine including PCV treatment).
3. Age 18 years or older.
4. Karnofsky performance status of 60 - 100 .
5. Not receiving another experimental treatment for glioblastoma at the moment of inclusion or during active treatment within the assigned group (i.e. control or disulfiram group).
6. Able to take oral medications.
7. No known allergy to disulfiram or copper.
8. Absolute neutrophil count ≥ 1,500/mcL and platelets ≥ 100,000/mcL
9. Serum/plasma copper and serum ceruloplasmin within institutional limits.

   a. However increased levels are seen together with ongoing acute phase reaction as determined by elevated C-reactive protein (ceruloplasmin is elevated as part of the same process) it is possible to retest after normalization of C-reactive protein.
10. Willing to refrain from ingestion of alcoholic beverages while on the study is a criteria to be randomized. However, once randomized alcohol abstinence only affects the group treated with disulfiram, and in this group it includes the entire period and one month after last dosage of disulfiram.

Exclusion Criteria:

1. Earlier treatment for progression (e.g. "rescue therapy")
2. History of idiopathic seizure disorder, psychosis or schizophrenia.
3. History of uncontrolled hypertension (i.e. systolic BP > 180 mmHg) and a diagnosis of congestive heart failure
4. Received radiotherapy within the 3 months before the diagnosis of progression .
5. Addiction to alcohol or drugs.
6. Pregnant and/or breastfeeding.
7. Women of childbearing potential who do not have negative pregnancy test not older than 14 days before enrollment.
8. History of active liver disease, including chronic active hepatitis, viral hepatitis (hepatitis B, C and CMV), cholestatic jaundice of any etiology or toxic hepatitis or inadequate hepatic function, defined as baseline ASAT and ALAT > 2.5 X upper institutional limit and/or bilirubin > 2.0 X upper institutional limit.
9. History of Wilson's disease or family member with Wilson's disease (unless excluded as a carrier by genetic test).
10. History of hemochromatosis or family member with hemochromatosis (unless excluded as a carrier by genetic test).
11. Nickel hypersensitivity (disulfiram mobilize nickel causing a brief increase in nickel concentrations before excretion. The initial increase may lead to hepatitis and predisposed patients).
12. Need for metronidazole, warfarin and/or theophylline medication (the metabolism may be influenced by disulfiram).
13. Patients who are taking medications metabolized by cytochrome P450 2E1, including chlorzoxazone or halothane and its derivatives (phenytoin, phenobarbital, chlordiazepoxide, imipramine, diazepam, isoniazid, metronidazole, warfarin, amitriptyline within 14 days prior to the first dose of disulfiram. Of note, lorazepam and oxazepam are not affected by the P450 system and are not contraindicated with disulfiram).
14. Unfit for participation for any other reason judged by the including physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-01; Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Survival 6 mo | Proportion of alive participants at 6 months

SECONDARY OUTCOMES:
Progression free survival | Proportion without progression at 6 and 12 months
  Using RANO criteria applied by local investigators
Survival 12 and 24 mo | Proportion of alive participants at 12 and 24 months
Median overall survival | Median overall survival assessed at 6 months and 24 months after last included participant
  Using Kaplan Meier plots and log-rank test
Health related quality of life | Assessed at baseline and month 3, 6, 9, 12, 15, 18, 21, 24
  EuroQol 5D (generic)
Volumetric tumor assessment | Baseline and first follow-up scan being scheduled at 3 months post-inclusion
  Tumor volumes are assessed using semi-automatic segmentation
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Assessed month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 15, 18, 21, 24, but analyzed as cumulative burden at 6 and 24 months
  Cumulative burden at 6 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir S Jakola, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (8):
- Cancer Clinic, St.Olavs University Hospital, Trondheim, Norway
- Sweden (7):
  - Dept. of Oncology, Sahlgrenska University Hospital, Gothenburg
  - Ryhov County Hospital, Jönköping
  - Linköping University Hospital, Linköping
  - Lund University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cvek B. Targeting malignancies with disulfiram (Antabuse): multidrug resistance, angiogenesis, and proteasome. Curr Cancer Drug Targets. 2011 Mar;11(3):332-7. doi: 10.2174/156800911794519806. PMID 21247389
- [Background] Nechushtan H, Hamamreh Y, Nidal S, Gotfried M, Baron A, Shalev YI, Nisman B, Peretz T, Peylan-Ramu N. A phase IIb trial assessing the addition of disulfiram to chemotherapy for the treatment of metastatic non-small cell lung cancer. Oncologist. 2015 Apr;20(4):366-7. doi: 10.1634/theoncologist.2014-0424. Epub 2015 Mar 16. PMID 25777347
- [Background] Triscott J, Rose Pambid M, Dunn SE. Concise review: bullseye: targeting cancer stem cells to improve the treatment of gliomas by repurposing disulfiram. Stem Cells. 2015 Apr;33(4):1042-6. doi: 10.1002/stem.1956. PMID 25588723
- [Background] Wickstrom M, Danielsson K, Rickardson L, Gullbo J, Nygren P, Isaksson A, Larsson R, Lovborg H. Pharmacological profiling of disulfiram using human tumor cell lines and human tumor cells from patients. Biochem Pharmacol. 2007 Jan 1;73(1):25-33. doi: 10.1016/j.bcp.2006.08.016. Epub 2006 Aug 26. PMID 17026967
- [Background] Dufour P, Lang JM, Giron C, Duclos B, Haehnel P, Jaeck D, Jung JM, Oberling F. Sodium dithiocarb as adjuvant immunotherapy for high risk breast cancer: a randomized study. Biotherapy. 1993;6(1):9-12. doi: 10.1007/BF01877380. PMID 8389572
- [Derived] Werlenius K, Kinhult S, Solheim TS, Magelssen H, Lofgren D, Mudaisi M, Hylin S, Bartek J Jr, Strandeus M, Lindskog M, Rashid HB, Carstam L, Gulati S, Solheim O, Bartek J, Salvesen O, Jakola AS. Effect of Disulfiram and Copper Plus Chemotherapy vs Chemotherapy Alone on Survival in Patients With Recurrent Glioblastoma: A Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e234149. doi: 10.1001/jamanetworkopen.2023.4149. PMID 37000452
- [Derived] Jakola AS, Werlenius K, Mudaisi M, Hylin S, Kinhult S, Bartek J Jr, Salvesen O, Carlsen SM, Strandeus M, Lindskog M, Lofgren D, Rydenhag B, Carstam L, Gulati S, Solheim O, Bartek J, Solheim T. Disulfiram repurposing combined with nutritional copper supplement as add-on to chemotherapy in recurrent glioblastoma (DIRECT): Study protocol for a randomized controlled trial. F1000Res. 2018 Nov 15;7:1797. doi: 10.12688/f1000research.16786.1. eCollection 2018. PMID 30647912